CLINICAL TRIAL: NCT06455072
Title: Nituzumab Plus Serplulimab Combined With SBRT in Recurrent Advanced Cervical Cancer: A Prospective, Multicenter, Single-arm, Phase II Clinical Trial
Brief Title: Nituzumab Plus Serplulimab Combined With SBRT in Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2022173
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Antibodies, Monoclonal; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nituzumab Plus Serplulimab Combined With SBRT (Experimental): Nituzumab was given intravenously (400mg qw, 21 days per cycle), and Serplulimab was administered intravenously (200mg once every 3 weeks).The dose was 30-50 Gy in three to five fractions and the number of lesions was no more than four by SBRT. The treatment was continued until disease progression, death or intolerant toxicity.
  Interventions: Drug: Nituzumab; Drug: Serplulimab

INTERVENTIONS:
Drug: Nituzumab — EGFR monoclonal antibody
  Other Names: monoclonal antibody
Drug: Serplulimab — PD-1 (programmed death receptor 1) monoclonal antibody
  Other Names: Immune checkpoint inhibitors

SUMMARY:
In recurrent advanced cervical cancer, patients were prone to drug resistance who have relapsed within prior platinum-based chemotherapy. However, immune checkpoint inhibitor's combination therapy has become a promising strategy for advanced cervical cancer. Epidermal Growth Factor Receptor (EGFR) is overexpressed in cervical cancer cells. Stereotactic radiotherapy (SBRT) can enhance the efficacy of immunotherapy.

DETAILED DESCRIPTION:
In recurrent advanced cervical cancer, patients were prone to drug resistance who have relapsed within prior platinum-based chemotherapy. However, immune checkpoint inhibitor's combination therapy has become a promising strategy for advanced cervical cancer. Epidermal Growth Factor Receptor (EGFR) is overexpressed in cervical cancer cells. Stereotactic radiotherapy (SBRT) can enhance the efficacy of immunotherapy.

Nituzumab is a humanized monoclonal antibody that binds to the epidermal growth factor receptor. Serplulimab is a fully humanized, high-affinity monoclonal antibody against programmed cell death-1 (PD-1).

This phase II, single-arm study aims to evaluate the efficacy and safety of Nituzumab plus Serplulimab combined with SBRT in patients with recurrent advanced cervical cancer.

Patients who have failed in standard chemotherapy，histopathologically confirmed recurrent advanced squamous cell cervical carcinoma regardless of programmed cell death-Ligand 1 (PD-L1) expression. Patients who have achieved the response state or come to stably at least six months after immunotherapy were allowed. There was at least one lesion for SBRT in addition to target lesions. ECOG 0-1 were considered eligible for enrollment.

Nituzumab was given intravenously (400mg qw, 21 days per cycle), and Serplulimab was administered intravenously (200mg once every 3 weeks).The dose was 30-50 Gy in three to five fractions and the number of lesions was no more than four by SBRT. The treatment was continued until disease progression, death or intolerant toxicity.

The primary endpoint was objective response rate (ORR) and the secondary endpoints included disease control rate (DCR), progression free survival (PFS), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1) Prospective participants will be voluntarily enrolled in this research study and will provide written informed consent, demonstrating the ability to adhere to scheduled visits and associated procedures.

  2) Individuals aged between 18 and 75 years old are eligible for inclusion. 3) Patients with histologically or cytologically confirmed cervical squamous cell carcinoma, along with documented disease progression that is unresponsive to curative treatment. It should be noted that confirmation of the original primary tumor tissue by a pathological report is required.

  4) Ineligibility due to failure of standard systemic treatment for persistent, recurrent, or metastatic cervical cancer (defined as progression or recurrence within six months after at least one cycle of standard systemic treatment; patients who have previously received anti-PD-1/PD-L1 antibody treatment and achieved CR, PR, or SD≥6 months may still be considered).

  5) Not suitable for local treatments such as curative surgery or radiotherapy. 6) A minimum interval of four weeks must occur between the completion of prior systemic therapy and administration of the investigational drug. Additionally, any treatment-related adverse events must have resolved to CTCAE V5.0 grade ≤1 (excluding hair loss and fatigue).

  7) At least one measurable lesion must serve as a target lesion according to RECIST V1.1 criteria.

  8) Presence of at least one non-target lesion amenable to SBRT is also necessary.

  9) Eastern Cooperative Oncology Group Performance Status (ECOG PS) score should be either 0 or 1.

  10）Expected survival time should exceed 12 weeks 11）Female subjects capable of reproduction need to utilize effective contraception throughout the study period and for at least five months following their final dose of the investigational drug 12）Subjects are required to consent providing sufficient tumor tissue samples for EGFR expression detection including archived tumor samples (paraffin blocks or an adequate number of unstained slides meeting study requirements); if no archived tumor tissue samples are available, subjects must agree on biopsy from the tumor site 13）Good organ function and bone marrow hematopoietic function.

Exclusion Criteria:

1. Diagnosed with malignancies other than basal cell carcinoma, squamous cell carcinoma of the skin, in situ carcinoma cured by surgical resection, and/or papillary thyroid carcinoma cured by surgery within 5 years prior to the initial dose. Participants must have pathological types other than cervical squamous cell carcinoma.
2. Participants presenting with clinical symptoms or requiring drainage due to pleural effusion, ascites, or pericardial effusion are eligible for inclusion, except those whose effusion does not require drainage or ceases draining within 3 days without a significant increase.
3. Participants who are scheduled for or have previously undergone organ or bone marrow transplantation.
4. Individuals with acute or chronic active hepatitis B or C infection, who have HBV DNA levels greater than 200IU/ml or 103 copies/ml, or are positive for anti-HCV antibodies with HCV-RNA levels above the detection limit may be eligible. Additionally, individuals with acute or chronic active hepatitis B or C infection who have been treated with nucleoside analog antiviral agents and have HBV DNA or HCV-RNA levels below the specified criteria or below the detection limit may also be eligible.
5. Individuals with meningeal metastasis or symptomatic central nervous system (CNS) metastasis may be considered for this study. Furthermore, individuals with asymptomatic brain metastasis that has been treated and symptoms stabilized for at least 2 weeks may also qualify if they meet specific criteria: presence of measurable lesions outside of the CNS; absence of metastasis to certain areas within the brain; no history of intracranial hemorrhage; discontinuation of hormone therapy at least 14 days prior to receiving the first dose of study drug.
6. Any life-threatening bleeding event within the past 3 months, including the requirement for blood transfusion, surgical intervention or local treatment, or ongoing pharmacological therapy.
7. Any arterial thrombosis, embolism, or ischemia within the past 6 months, such as myocardial infarction, unstable angina, or cerebrovascular accident. A history of any significant thromboembolic event within the past 3 months, such as deep vein thrombosis or any other thromboembolic event (thrombosis related to a portacatheter or central venous catheter insertion site, superficial vein thrombosis, or a stable post-treatment thrombosis is not considered "significant" thromboembolic event).
8. Hepatic vein thrombus involving both the hepatic trunk and the left and right branches, or involving both the trunk and the superior mesenteric vein, inferior vena cava; superior vena cava thrombus, superior vena cava syndrome.
9. Tumor invasion of surrounding important organs or blood vessels (such as the great vessels of the mediastinum, the superior vena cava, the inferior vena cava, the abdominal aorta, the iliac vessels, the trachea, the esophagus, etc.), or the risk of developing a tracheo-esophageal fistula or an esophago-pleural fistula.
10. Uncontrollable hypertension, with a systolic blood pressure of ≥150mmHg or a diastolic blood pressure of ≥100mmHg, history of hypertension crisis or hypertension cerebral infarction.
11. Symptomatic congestive heart failure (New York Heart Association classification II-IV). Symptomatic or uncontrolled arrhythmia. QT interval prolongation, QTcF>470ms.
12. Severe bleeding tendency or coagulation disorder, or currently receiving thrombolytic therapy.
13. History of gastrointestinal perforation and/or fistula within the past 6 months, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive bowel resection (partial colon resection or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
14. History of interstitial pneumonitis, drug-induced pneumonitis, radiation pneumonitis, idiopathic pneumonitis, or active pneumonitis. 15) Active tuberculosis (TB), who are currently receiving anti-TB treatment or have received anti-TB treatment within 1 year prior to the start of the study.

16) Individuals with Human Immunodeficiency Virus (HIV) infection (HIV 1/2 antibody positive), known active syphilis infection.

17) Severe infections that are active or not well controlled. A severe infection within 4 weeks prior to the first dose, including but not limited to hospitalization due to infection, sepsis, or severe pneumonia complications.

18) Oral or intravenous administration of therapeutic antibiotics within 1 week prior to the start of the study.

19) Active systemic autoimmune diseases or a history of such disease within the past 2 years (Psoriasis, alopecia, vitiligo, or Graves' disease that do not require systemic treatment within the past 2 years, hypothyroidism that only requires thyroid hormone replacement therapy, and type 1 diabetes that only requires insulin replacement therapy can be included). A history of primary immunodeficiency is known. Only individuals with positive autoimmune antibodies need to be confirmed by the investigator for the presence of autoimmune diseases. 20) You have used an immunosuppressive drug within the past 4 weeks, excluding topical or inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e., no more than 10 mg of prednisone or equivalent daily doses of other corticosteroids) used for the relief of breathing difficulties associated with conditions such as asthma or chronic obstructive pulmonary disease.

21) You have received a live attenuated vaccine within the past 4 weeks or plan to receive one during the study.

22) You have received systemic immune stimulation therapy within the past 4 weeks.

23) You have had a major surgical procedure (craniotomy, thoracotomy, or laparotomy) within the past 4 weeks or have an unhealed wound, ulcer, or fracture.

24) You have an uncontrolled/uncorrectable metabolic disorder or other non-malignant tumor organ disease or systemic disease or cancer-related complications that may result in higher medical risk and/or uncertainty in survival assessment.

25) You have any other acute or chronic disease, mental illness, or laboratory test abnormality that may increase the risk of participating in the study or receiving study medication, or interfere with the interpretation of study results, as determined by the investigator.

26) You have previously received nintedanib or other anti-EGFR therapy. 27) You have previously received sunitinib therapy. 28) Previous treatment with anti-CTLA-4 antibody.

29) Known to be allergic to any nivolumab, siltuximab component; or had a severe allergic reaction to other monoclonal antibodies in the past.

30) Received any anti-cancer treatment within 4 weeks prior to starting the study: systemic chemotherapy (oral fluoropyrimidine washout period is 2 weeks), endocrine therapy, targeted therapy (small molecule targeted therapy washout period is 2 weeks or 5.5 half-lives, whichever is longer), immunotherapy, tumor embolization therapy, or traditional Chinese medicine treatment for anti-cancer indications, etc.

31）Pregnant or breastfeeding female patients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 2years
  objective response rate

SECONDARY OUTCOMES:
PFS | 2years
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Qin Xu, Study Director — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China